CLINICAL TRIAL: NCT01366638
Title: A Phase III, Open-Label Study in Japan to Assess the Efficacy and Safety of TMC435 as Part of a Treatment Regimen Including Peginterferon Alfa-2b and Ribavirin in Hepatitis C, Genotype 1 Infected Subjects
Brief Title: A Study of TMC435 in Participants With Genotype 1 Hepatitis C Virus (HCV) Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR017935; TMC435HPC3010 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2011-06-02; First posted 2011-06-06 (Estimated); Results first posted 2014-01-20 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-04

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C, Chronic; TMC435; Hepatitis C; Hepatitis C virus; Interferon Alfa-2b; Ribavirin; Viral ribonucleic acid
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — Simeprevir; peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment-Naive: TMC435 100 mg 12 Wks+PR 24/48 (Experimental): Participants will receive TMC435 100 mg once daily with PegIFNa-2b and ribavirin (PR) for 12 weeks (Wks), followed by PR until Week 24 or Week 48. Treatment will be stopped at Week 24 in participants who achieve plasma hepatitis C virus (HCV) ribonucleic acid (RNA) levels <1.2 log10 IU/mL detectable or undetectable at Week 4, and undetectable plasma HCV RNA levels at Week 12. All other participants will continue PR until Week 48.
  Interventions: Drug: TMC435; Drug: Peginterferon alfa-2b (pegIFN alfa-2b); Drug: Ribavirin (RBV)
- Prior Relapser: TMC435 100 mg 12 Wks+PR 24/48 (Experimental): Participants will receive TMC435 100 mg once daily with PegIFNa-2b and ribavirin (PR) for 12 weeks (Wks) followed by PR until Week 24. Treatment will be stopped at Week 24 in participants who achieve plasma hepatitis C virus (HCV) ribonucleic acid (RNA) levels <1.2 log10 IU/mL detectable or undetectable at Week 4, and undetectable plasma HCV RNA levels at Week 12. All other participants will continue PR until Week 48.
  Interventions: Drug: TMC435; Drug: Peginterferon alfa-2b (pegIFN alfa-2b); Drug: Ribavirin (RBV)
- Prior Non-Responder: TMC435 100 mg 12 Wks+PR 48 (Experimental): Participants will receive TMC435 100 mg once daily with PegIFNa-2b and ribavirin (PR) for 12 weeks (Wks) followed by PR until Week 48.
  Interventions: Drug: TMC435; Drug: Peginterferon alfa-2b (pegIFN alfa-2b); Drug: Ribavirin (RBV)

INTERVENTIONS:
Drug: TMC435 — 100 mg capsule taken by mouth once daily for 12 weeks
Drug: Peginterferon alfa-2b (pegIFN alfa-2b) — PegIFN alfa-2b will be supplied as a vial containing dried and frozen powder with 74,148 or 222 mcg pegIFN alpha-2b attached to 0.7 ml injection water (50, 100 or 150 mcg/0.5mL pegIFN alpha-2b) and will be administered according to the manufacturer's prescribing information as 1.5 mcg/kg once weekly injected subcutaneous (under the skin) for up to 24-48 weeks.
  Other Names: PEGINTRON
Drug: Ribavirin (RBV) — The dose of RBV given will be based on body weight. If body weight is > 80 kg the total daily dose of RBV will be 1000 mg, taken by mouth as 400 mg (2 capsules of 200 mg) after breakfast and 600 mg (3 capsules of 200 mg) after supper. If body weight is > 60 kg to <=80 kg the total daily dose will be 800 mg, taken by mouth as 400 mg (2 capsules of 200 mg per intake) after breakfast and supper. If body weight is <=60 kg the total daily dose of RBV will be 600 mg, taken by mouth as 200 mg (1 capsule of 200 mg) after breakfast and 400 mg (2 capsules of 200 mg) after supper. Total duration of RBV will be 24-48 weeks.
  Other Names: REBETOL

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of TMC435 in combination with peginterferon alfa-2b and ribavirin in chronic genotype 1 hepatitis C virus (HCV)-infected participants who are treatment-naive or treatment-experienced (prior relapser or non-responder to Interferon-based therapy) in Japan.

DETAILED DESCRIPTION:
This is an open-label study (all people involved know the identity of the intervention) to evaluate the efficacy and safety of TMC435 (also referred to as jnj-38733214-aaa) in combination with the standard of care therapy (SoC: peginterferon [pegIFN] alfa-2b and ribavirin) in adult, genotype 1 hepatitis C virus (HCV)-infected participants who are treatment-naive (never received treatment for HCV), prior relapsers (relapsed after previous interferon [IFN]-based therapy), or non-responders (failed to respond to previous IFN-based therapy) in Japan. The study objective is to evaluate the efficacy, safety, and pharmacokinetics of TMC435. A sufficient number of participants who are treatment-naive, prior relapsers to treatment with IFN-based therapy, and prior non-responders to treatment with IFN-based therapy will be enrolled and assigned to 1 of 3 panels (referred to as treatment groups). Participants who are treatment-naive or prior relapsers to IFN-based therapy will receive 12 weeks of treatment with TMC435 (100 mg) once daily with pegIFN alfa-2b and ribavirin (PR) followed by an additional 12 or 24 weeks of treatment with PR. Participants who are non-responders to IFN-based therapy will receive 12 weeks of treatment with TMC435 (100 mg) once daily with PR followed by an additional 36 weeks of treatment with PR. TMC435 is a 100-mg capsule and will be taken orally by mouth. The SoC treatment will consist of Pegylated interferon (PegIFN alpha-2b) (1.5 mcg/kg) injected with a syringe subcutaneously (under the skin) once weekly and ribavirin 200-mg capsules (daily dose: 600-1000 mg based on body weight) taken orally by mouth 2 times a day after meals for 24 or 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have chronic genotype 1 HCV infection with HCV RNA level >= 5.0 log10 IU/mL
* Patient has never received treatment for HCV (treatment-naive), relapsed after previous IFN-based therapy (prior relapser) or failed to respond to previous IFN-based therapy (non-responder)
* Patient must be willing to use contraceptive measures from the time of informed consent to 6 months after last dose of study medication.

Exclusion Criteria:

* Co-infection with any other HCV genotype or co-infection with the human immunodeficiency virus (HIV)
* Diagnosed with hepatic cirrhosis or hepatic failure
* A medical condition which is a contraindication to peg-IFN or ribavirin therapy
* History of, or any current medical condition, which could impact the safety of the patient in the study

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2011-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K. Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (11):
- Japan (11):
  - Amagasaki
  - Ikeda
  - Kawasaki
  - Kumamoto
  - Niigata
  - Ohmura
  - Osaka
  - Sakai
  - Sapporo
  - Suita
  - Tokyo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 01-Apr-2011 to 20-Nov-2012 and recruited participants with chronic Hepatitis C Virus (HCV) infection from 14 study centers in Japan. A total of 79 participants with chronic genotype 1 HCV infection were randomized and started treatment; 65 completed the study.
Pre-assignment Details: Participants with genotype 1 hepatitis C virus (HCV) infection who were treatment-naïve or treatment-experienced (prior relapsers or nonresponders to interferon-based therapy) were assigned to 1 of 3 groups and received TMC435 100 mg/day for 12 weeks coadministered with PegIFNa-2b + ribavirin until Week 24 or Week 48.
Groups:
- Treatment-Naive: TMC435 100 mg 12 Wks+PR 24/48: Participants received TMC435 100 mg once daily with PegIFNa-2b and ribavirin (PR) for 12 weeks (Wks), followed by PR until Week 24 or Week 48. Treatment was to be stopped at Week 24 in participants who achieved plasma hepatitis C virus (HCV) ribonucleic acid (RNA) levels <1.2 log10 IU/mL detectable or undetectable at Week 4, and undetectable plasma HCV RNA levels at Week 12. All other participants continued PR until Week 48.
- Prior Relapser: TMC435 100 mg 12 Wks+PR 24/48: Participants received TMC435 100 mg once daily with PegIFNa-2b and ribavirin (PR) for 12 weeks (Wks) followed by PR until Week 24. Treatment was to be stopped at Week 24 in participants who achieved plasma hepatitis C virus (HCV) ribonucleic acid (RNA) levels <1.2 log10 IU/mL detectable or undetectable at Week 4, and undetectable plasma HCV RNA levels at Week 12. All other participants continued PR until Week 48.
- Prior Non-Responder: TMC435 100 mg 12 Wks+PR 48: Participants received TMC435 100 mg once daily with PegIFNa-2b and ribavirin (PR) for 12 weeks (Wks) followed by PR until Week 48.
Period: Overall Study
Arm/Group | Treatment-Naive: TMC435 100 mg 12 Wks+PR 24/48 | Prior Relapser: TMC435 100 mg 12 Wks+PR 24/48 | Prior Non-Responder: TMC435 100 mg 12 Wks+PR 48
Started | 24 | 29 | 26
Completed | 23 | 29 | 20
Not Completed | 1 | 0 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 6
Not completed — Other | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment-Naive: TMC435 100 mg 12 Wks+PR 24/48 | Prior Relapser: TMC435 100 mg 12 Wks+PR 24/48 | Prior Non-Responder: TMC435 100 mg 12 Wks+PR 48 | Total
Number analyzed (Participants) | 24 | 29 | 26 | 79
Age, Continuous [Median (Full Range); unit: years] | 60 [37 to 68] | 60 [38 to 70] | 53 [45 to 69] | 60 [37 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 13 | 42
  Male | 8 | 16 | 13 | 37

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants With a Sustained Virologic Response 12 Weeks After the Actual End of Treatment (SVR12)
Description: The table below shows the percentage of participants in each treatment group with an SVR12 defined as participants with undetectable plasma Hepatitis C virus (HCV) ribonucleic acid (RNA) at the end of treatment (Week 24 or 48) who also had undetectable plasma HCV RNA 12 weeks after the last dose of treatment (Week 36 or 60). NOTE: All outcome measures reported in this study are "Exploratory;" not "Primary" as indicated (refer to Limits and Caveats).
Time Frame: Week 36 or 60
Population: The Full Analysis Set (FAS) consisted of all participants who received at least one dose of study drug during the study except for those who did not meet the major eligibility criteria for the study and participants who did not have efficacy data available after treatment with study medication.
Measure: Number; unit: Percentage of Participants
Arm/Group | Treatment-Naive: TMC435 100 mg 12 Wks+PR 24/48 | Prior Relapser: TMC435 100 mg 12 Wks+PR 24/48 | Prior Non-Responder: TMC435 100 mg 12 Wks+PR 48
Number analyzed (Participants) | 24 | 29 | 26
Percentage of Participants | 91.7 | 100.0 | 38.5

2. Primary Outcome: The Percentage of Participants With a Sustained Virologic Response 24 Weeks After the Actual End of Treatment (SVR24)
Description: The table below shows the percentage of participants in each treatment group with a SVR24 defined as participants with undetectable plasma hepatitis C virus (HCV) ribonucleic acid (RNA) at the end of treatment and at 24 weeks after the last dose of treatment (Week 48 or 72). NOTE: All outcome measures reported in this study are "Exploratory;" not "Primary" as indicated (refer to Limits and Caveats).
Time Frame: 24 weeks after the last dose of treatment (Week 48 or 72)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment-Naive: TMC435 100 mg 12 Wks+PR 24/48 | Prior Relapser: TMC435 100 mg 12 Wks+PR 24/48 | Prior Non-Responder: TMC435 100 mg 12 Wks+PR 48
Number analyzed (Participants) | 24 | 29 | 26
Percentage of participants | 91.7 | 96.6 | 38.5

3. Primary Outcome: The Percentage of Participants With Undetectable Plasma Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) During Treatment and at the End of Treatment
Description: The table below shows the percentage of participants in each treatment group with undetectable HCV RNA less than 1.2 log10 IU/mL during treatment and at end of treatment (EOT). NOTE: All outcome measures reported in this study are "Exploratory;" not "Primary" as indicated (refer to Limits and Caveats).
Time Frame: Weeks 4, 12, 24, 36, 48, 60, 72, and EOT (up to Week 48)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment-Naive: TMC435 100 mg 12 Wks+PR 24/48 | Prior Relapser: TMC435 100 mg 12 Wks+PR 24/48 | Prior Non-Responder: TMC435 100 mg 12 Wks+PR 48
Number analyzed (Participants) | 24 | 29 | 26
Percentage of participants
  Week 4 | 79.2 | 86.2 | 57.7
  Week 12 | 100 | 100 | 76.9
  Week 24 | 100 | 96.6 | 65.4
  Week 36 | 87.5 | 96.6 | 57.7
  Week 48 | 83.3 | 96.6 | 53.8
  Week 60 | 91.7 | 96.6 | 38.5
  Week 72 | 91.7 | 96.6 | 38.5
  EOT | 100 | 100 | 57.7

4. Primary Outcome: The Number of Participants With Viral Breakthrough
Description: The table below shows the number of participants in each treatment group who experienced viral breakthrough during the TMC435 treatment period. Viral breakthrough is defined as a confirmed increase of greater than 1 log10 IU/mL in plasma hepatitis C virus (HCV) ribonucleic acid (RNA) level from the lowest level reached or a confirmed value of plasma HCV RNA of greater than 2.0 log10 IU/mL in participants whose plasma HCV RNA level had previously been reported below 1.2 log10 IU/mL detectable or undetectable. NOTE: All outcome measures reported in this study are "Exploratory;" not "Primary" as indicated (refer to Limits and Caveats).
Time Frame: Up to 48 Weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Treatment-Naive: TMC435 100 mg 12 Wks+PR 24/48 | Prior Relapser: TMC435 100 mg 12 Wks+PR 24/48 | Prior Non-Responder: TMC435 100 mg 12 Wks+PR 48
Number analyzed (Participants) | 24 | 29 | 26
Participants | 0 | 0 | 2

5. Primary Outcome: The Number of Participants Demonstrating Viral Relapse
Description: The table below shows the number of participants in each treatment group who demonstrated viral relapse, defined as having undetectable plasma hepatitis C virus (HCV) ribonucleic acid (RNA) levels at end of treatment (EOT [Week 24 or 48]) and detectable HCV RNA during follow-up or detectable HCV RNA at the time points of an assessment of sustained virologic response (SVR). The number of participants analyzed in each treatment group below are those with undetectable HCV RNA levels at EOT and with at least one follow-up HCV RNA measurement. NOTE: All outcome measures reported in this study are "Exploratory;" not "Primary" as indicated (refer to Limits and Caveats).
Time Frame: Up to 72 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Treatment-Naive: TMC435 100 mg 12 Wks+PR 24/48 | Prior Relapser: TMC435 100 mg 12 Wks+PR 24/48 | Prior Non-Responder: TMC435 100 mg 12 Wks+PR 48
Number analyzed (Participants) | 24 | 29 | 15
Participants | 2 | 1 | 4

6. Primary Outcome: The Number of Participants With Abnormal Alanine Aminotransferase (ALT) Levels at Baseline Who Achieved Normal Limit of ALT at the End of Treatment (EOT)
Description: The table below shows the number of participants in each treatment group with abnormal ALT levels at Baseline who achieved normalization of ALT levels defined as having an ALT value less than or equal to the Upper Limit of Normality (ie, 40 IU/mL) at EOT. At Baseline, 15 treatment-naïve participants, 13 prior relapsers, and 13 prior non-responders had abnormal ALT levels at Baseline. NOTE: All outcome measures reported in this study are "Exploratory;" not "Primary" as indicated (refer to Limits and Caveats).
Time Frame: Up to Week 48
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment-Naive: TMC435 100 mg 12 Wks+PR 24/48 | Prior Relapser: TMC435 100 mg 12 Wks+PR 24/48 | Prior Non-Responder: TMC435 100 mg 12 Wks+PR 48
Number analyzed (Participants) | 15 | 13 | 13
Percentage of participants | 13 | 8 | 8

7. Primary Outcome: The Percentage of Participants Who Achieved a Greater Than or Equal to 2 log10 IU/mL Drop From Baseline in Plasma Hepatitis C Virus Ribonucleic Acid (HCV RNA) at Each Time Point During Treatment and Follow-up
Description: The table below shows the percentage of participants in each treatment group with greater than or equal to 2 log10 IU/mL drop from baseline in plasma hepatitis C virus (HCV) ribonucleic acid (RNA) at each time point during treatment and post-treatment follow-up. NOTE: All outcome measures reported in this study are "Exploratory;" not "Primary" as indicated (refer to Limits and Caveats).
Time Frame: Day 3, Day 7 and Weeks 2, 3, 4, 8, 12, 16, 20, 24, 28, 36, 48, 60, 72, EOT (up to Week 24 or 48), follow-up (FU) Week 4, 12, and 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment-Naive: TMC435 100 mg 12 Wks+PR 24/48 | Prior Relapser: TMC435 100 mg 12 Wks+PR 24/48 | Prior Non-Responder: TMC435 100 mg 12 Wks+PR 48
Number analyzed (Participants) | 24 | 29 | 26
Percentage of participants
  Day 3 | 100 | 100 | 88.5
  Day 7 | 100 | 100 | 100
  Week 2 | 100 | 100 | 100
  Week 3 | 100 | 100 | 96.2
  Week 4 | 100 | 100 | 96.2
  Week 8 | 100 | 100 | 92.3
  Week 12 | 100 | 100 | 84.6
  Week 16 | 100 | 96.6 | 76.9
  Week 20 | 95.8 | 100 | 76.9
  Week 24 | 100 | 96.6 | 73.1
  Week 28 | 91.7 | 96.6 | 69.2
  Week 36 | 87.5 | 96.6 | 65.4
  Week 48 | 83.3 | 96.6 | 61.5
  Week 60 | 91.7 | 96.6 | 42.3
  Week 72 | 91.7 | 96.6 | 38.5
  EOT | 100 | 100 | 80.8
  FU Week 4 | 95.8 | 100 | 46.2
  FU Week 12 | 91.7 | 100 | 42.3
  FU Week 24 | 91.7 | 96.6 | 38.5

8. Primary Outcome: The Percentage of Participants Who Met Response Guided Treatment (RGT) Criteria and Completed Treatment With Peginterferon Alpha-2b (PegIFNα-2b) and Ribavirin (RBV) at Week 24
Description: The table below shows the percentage of participants in each treatment group who met RGT criteria (ie, who had plasma levels of hepatitis C virus ribonucleic acid [HCV RNA] <1.2 log10 IU/mL detectable/undetectable at Week 4 and <1.2 log 10 IU/mL undetectable at Week 12) and completed treatment with PegIFNα-2b and RBV at Week 24. Participants in the TMC435 Treatment-Naïve and TMC435 Prior Relapser treatment groups not meeting RGT criteria continued treatment with PegIFNα-2a and RBV to Week 48 (does not apply to the TMC435 Non-responder treatment group because the specified treatment duration was 48 weeks and RGT criteria was not assessed at Week 24). NOTE: All outcome measures reported in this study are "Exploratory;" not "Primary" as indicated (refer to Limits and Caveats).
Time Frame: Week 24 or 48
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment-Naive: TMC435 100 mg 12 Wks+PR 24/48 | Prior Relapser: TMC435 100 mg 12 Wks+PR 24/48
Number analyzed (Participants) | 24 | 29
Percentage of participants | 91.7 | 96.6

9. Primary Outcome: The Area Under the Plasma Concentration-Time Curve (From 0 to 24 Hours) (AUC24h)
Description: The table below shows the median (range) AUC24h values for TMC435 for all participants in each TMC435 treatment group who received TMC435 for up to 12 weeks. "Overall" is the median exposure estimate using all available data for each participant in the study. NOTE: All outcome measures reported in this study are "Exploratory;" not "Primary" as indicated (refer to Limits and Caveats).
Time Frame: Overall (Up to Week 12)
Population: Pharmacokinetic (PK) analysis was performed in the PK population, defined as all participants from whom sparse blood samples were drawn and who received at least 1 dose of study medication.
Measure: Median (Full Range); unit: ng·h/mL
Arm/Group | Treatment-Naive: TMC435 100 mg 12 Wks+PR 24/48 | Prior Relapser: TMC435 100 mg 12 Wks+PR 24/48 | Prior Non-Responder: TMC435 100 mg 12 Wks+PR 48
Number analyzed (Participants) | 24 | 29 | 26
ng·h/mL | 35448 [17659 to 87904] | 68130 [22208 to 248340] | 40645 [18222 to 240055]

10. Primary Outcome: Plasma Concentrations of TMC435
Description: The table below shows the median (range) TMC435 predose plasma concentrations (C0h) and maximum concentration (Cmax) values for participants in each treatment group. "Overall" is the median exposure estimate using all available data for each participant in the study. NOTE: All outcome measures reported in this study are "Exploratory;" not "Primary" as indicated (refer to Limits and Caveats).
Time Frame: Overall (Up to Week 12)
Population: as for outcome 9
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Treatment-Naive: TMC435 100 mg 12 Wks+PR 24/48 | Prior Relapser: TMC435 100 mg 12 Wks+PR 24/48 | Prior Non-Responder: TMC435 100 mg 12 Wks+PR 48
Number analyzed (Participants) | 24 | 29 | 26
ng/mL
  Cmax | 2304 [1593 to 4450] | 3643 [1780 to 11117] | 2521 [1616 to 10776]
  C0h | 735 [171 to 2842] | 2015 [287 to 9520] | 921 [184 to 9167]

ADVERSE EVENTS:
Time Frame: Up to approximately 52 weeks (includes all serious and other adverse events that newly occurred or worsened after treatment with TMC435, PegIFNα-2b or ribavirin, until the end date of the last study medication intake + 28 days)
Arm/Group | Treatment-Naive: TMC435 100 mg 12 Wks+PR 24/48 | Prior Relapser: TMC435 100 mg 12 Wks+PR 24/48 | Prior Non-Responder: TMC435 100 mg 12 Wks+PR 48
Serious Adverse Events (participants affected / at risk) | 1/24 | 0/29 | 1/26
Other Adverse Events (participants affected / at risk) | 24/24 | 29/29 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment-Naive: TMC435 100 mg 12 Wks+PR 24/48 (N=24) | Prior Relapser: TMC435 100 mg 12 Wks+PR 24/48 (N=29) | Prior Non-Responder: TMC435 100 mg 12 Wks+PR 48 (N=26)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0
Peripheral T-cell lymphoma unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment-Naive: TMC435 100 mg 12 Wks+PR 24/48 (N=24) | Prior Relapser: TMC435 100 mg 12 Wks+PR 24/48 (N=29) | Prior Non-Responder: TMC435 100 mg 12 Wks+PR 48 (N=26)
Pyrexia (General disorders) | 18 | 27 | 22
Malaise (General disorders) | 12 | 12 | 14
Injection site reaction (General disorders) | 11 | 8 | 12
Fatigue (General disorders) | 6 | 7 | 1
Injection site erythema (General disorders) | 5 | 2 | 1
Chills (General disorders) | 2 | 1 | 1
White blood cell count decreased (Investigations) | 17 | 16 | 13
Neutrophil count decreased (Investigations) | 11 | 8 | 7
Platelet count decreased (Investigations) | 11 | 6 | 8
Haemoglobin decreased (Investigations) | 10 | 2 | 5
Haematocrit decreased (Investigations) | 8 | 2 | 1
Red blood cell count decreased (Investigations) | 7 | 2 | 1
Blood albumin decreased (Investigations) | 5 | 1 | 0
Blood bilirubin increased (Investigations) | 5 | 12 | 6
Blood calcium decreased (Investigations) | 5 | 1 | 1
Blood cholesterol decreased (Investigations) | 5 | 0 | 1
Lymphocyte percentage increased (Investigations) | 5 | 0 | 0
Bilirubin conjugated increased (Investigations) | 4 | 0 | 0
Blood bilirubin unconjugated increased (Investigations) | 4 | 0 | 0
Weight decreased (Investigations) | 4 | 3 | 3
Eosinophil percentage increased (Investigations) | 3 | 0 | 0
High density lipoprotein decreased (Investigations) | 3 | 0 | 0
Lipase increased (Investigations) | 3 | 4 | 0
Blood uric acid increased (Investigations) | 2 | 1 | 0
Monocyte percentage increased (Investigations) | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 2 | 0
Liver function test abnormal (Investigations) | 0 | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 14 | 9 | 5
Rash (Skin and subcutaneous tissue disorders) | 12 | 8 | 10
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 7 | 6
Erythema (Skin and subcutaneous tissue disorders) | 3 | 2 | 1
Heat rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 10 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 3 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 5 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 6 | 0 | 6
Stomatitis (Gastrointestinal disorders) | 6 | 6 | 9
Nausea (Gastrointestinal disorders) | 4 | 5 | 2
Abdominal discomfort (Gastrointestinal disorders) | 3 | 2 | 4
Constipation (Gastrointestinal disorders) | 3 | 1 | 0
Cheilitis (Gastrointestinal disorders) | 2 | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 2
Dental caries (Gastrointestinal disorders) | 0 | 1 | 3
Anaemia (Blood and lymphatic system disorders) | 11 | 21 | 8
Neutropenia (Blood and lymphatic system disorders) | 6 | 2 | 5
Leukopenia (Blood and lymphatic system disorders) | 4 | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 12 | 12 | 7
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 2
Headache (Nervous system disorders) | 11 | 12 | 13
Dysgeusia (Nervous system disorders) | 4 | 3 | 1
Somnolence (Nervous system disorders) | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Insomnia (Psychiatric disorders) | 4 | 4 | 7
Nasopharyngitis (Infections and infestations) | 3 | 7 | 6
Cystitis (Infections and infestations) | 1 | 1 | 2
Dry eye (Eye disorders) | 2 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 4 | 3
Hypertension (Vascular disorders) | 2 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 2 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 2

LIMITATIONS AND CAVEATS:
All outcome measures reported in this study are "Exploratory;" not "Primary" as indicated. "Primary" was chosen for each outcome measure because "Exploratory" is not available as an outcome measure type on this form.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.